CLINICAL TRIAL: NCT05918718
Title: Assessment of the Efficacy of Letrozole in Comparison to Methotrexate in the Treatment of Ectopic Pregnancy
Brief Title: Assessment of the Efficacy of Letrozole in the Treatment of Ectopic Pregnancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.TUMS.IKHC.REC.1401.093
Record Dates: First submitted 2023-04-08; First posted 2023-06-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-04

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Letrozole; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- methotrexate (Experimental): The first group will receive a single dose (50 mg/m2) of methotrexate The beta-hcg level is measured on the first day, and the hcg serum level is routinely measured on the fourth, seventh and fourteenth day.
  Interventions: Drug: methotrexate
- Letrozole BD (Experimental): The first group will receive letrozole is given in the form of 2.5 mg tablets twice a day for 10 days. And on the fourth, seventh and fourteenth day, the HCG level is measured.
  Interventions: Drug: Letrozole
- Letroozole TDS (Experimental): letrozole is given in the form of 2.5 mg tablets 3 times a day for 5 days, and hCG levels are measured on days 4, 7, and 14.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — assessment of the efficacy of Letrozole in treatment of ectopic pregnancy
  Arms: Letroozole TDS; Letrozole BD
Drug: methotrexate — methotrexate
  Arms: methotrexate

SUMMARY:
In this study, about 150 women diagnosed with ectopic pregnancy who are referred to the Obstetrics and Gynecology Center of Valiasr Hospital are included in the study. Demographic information including both gynecological and obstetrical data is collected. Ectopic ectopic pregnancy is confirmed by transvaginal ultrasound. The patients are randomly allocated to three groups The first group will receive a single dose of methotrexate The second group will receive letrozole within a 10-day period, twice a day The third group will receive letrozole in a 5-day period three times a day In the first group, the first day of drug injection is counted, and the drug is measured at a dose of 50 mg/m2 and divided intramuscularly. The hcg level is measured on the first day, and the hcg serum level is routinely measured on the fourth, seventh and fourteenth day.

In the second group, letrozole is given in the form of 2.5 mg tablets twice a day for 10 days. And on the fourth, seventh and fourteenth day, the HCG level is measured.

In the third group, letrozole is given in the form of 2.5 mg tablets 3 times a day for 5 days, and hCG levels are measured on days 4, 7, and 14.

Also, the level of blood cells, liver enzymes, urea level and serum creatinine level are measured on the first day and the seventh day after the treatment.

The level of antimullerin hormone is measured on the first day and 3 months after the treatment.

DETAILED DESCRIPTION:
In this study, about 150 women diagnosed with ectopic pregnancy who are referred to the Obstetrics and Gynecology Center of Valiasr Hospital are included in the study. Demographic information including both gynecological and obstetrical data is collected. Ectopic ectopic pregnancy is confirmed by transvaginal ultrasound. The patients are randomly allocated to three groups The first group will receive a single dose of methotrexate The second group will receive letrozole within a 10-day period, twice a day The third group will receive letrozole in a 5-day period three times a day In the first group, the first day of drug injection is counted, and the drug is measured at a dose of 50 mg/m2 and divided intramuscularly. The hcg level is measured on the first day, and the hcg serum level is routinely measured on the fourth, seventh and fourteenth day.

In the second group, letrozole is given in the form of 2.5 mg tablets twice a day for 10 days. And on the fourth, seventh and fourteenth day, the HCG level is measured.

In the third group, letrozole is given in the form of 2.5 mg tablets 3 times a day for 5 days, and hCG levels are measured on days 4, 7, and 14.

Also, the level of blood cells, liver enzymes, urea level and serum creatinine level are measured on the first day and the seventh day after the treatment.

The level of antimullerin hormone is measured on the first day and 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18-40 years of age who have spontaneously conceived and ectopic pregnancy has been definitively diagnosed.

Exclusion Criteria:

* B-HCG levels more or equal to 5000
* Hemoglobin level less than 10 g/dl Platelet level less than 100,000
* Increasing the level of liver function tests and the level of urea and creatinine The presence of fetal heart activity in the gestational sac

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
βhCG | on day 14
Anti mulerian hormone | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: azadeh tarafdari, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital Complex, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarafdari A, Eslami Khotbesara S, Keikha F, Parsaei M, Poorabdoli M, Chill HH, Hadizadeh A. Comparing the effectiveness of letrozole versus methotrexate for treatment of ectopic pregnancy: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2024 Aug;299:219-224. doi: 10.1016/j.ejogrb.2024.06.026. Epub 2024 Jun 17. PMID 38901084